CLINICAL TRIAL: NCT05337787
Title: Effects of the Flipped Learning Model on Blood Pressure Knowledge and Self-directed Learning Skills of First-Year Nursing Students: A Randomized Controlled Study
Brief Title: Flipped Classroom Approach on Nursing Students' Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Emel Gülnar, Assistant professor, Kırıkkale University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: NCT
Record Dates: First submitted 2022-04-07; First posted 2022-04-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Nursing Student; Blood Pressure; Education

STUDY DESIGN:
Who Masked: Participant
Masking Description: Students were divided into intervention and control groups by simple randomization method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The students in the experimental group were trained using the flipped learning model.
  Interventions: Other: flipped classroom approach
- Control (No Intervention): The students in the control group were trained using only a traditional education method.

INTERVENTIONS:
Other: flipped classroom approach — The students in the experimental group were trained using the flipped learning model.
  Arms: Experimental

SUMMARY:
Effects of the Flipped Learning Model on Blood Pressure Knowledge and Self-directed Learning Skills of First-Year Nursing Students: A Randomized Controlled Study

DETAILED DESCRIPTION:
This study is to determine the effect of flipped learning model on blood pressure knowledge level and self-directed learning skills of first-year nursing students.

This study was a pre-post test open-label randomized controlled trial. Settings and Participants: This research was conducted with 94 first-year students (experimental group = 48, control group = 46) studying at a university in Turkey, Faculty of Health Sciences, Department of Nursing. The students were divided into experimental and control groups using a simple randomization method. The study data were collected using the Descriptive Characteristics Form, the Blood Pressure Knowledge Test, and the Self-Managed Learning Skills Scale. The students in the experimental group were trained using the flipped learning model. The students in the control group were trained using only a traditional education method.

ELIGIBILITY:
Inclusion Criteria:

* The first to enroll in the Fundamentals of Nursing course,
* Volunteer to participate in the research
* had continuous Internet Access

Exclusion Criteria:

* Having graduated from Health Vocational High School or having studied a health-related department,
* Have taken fundamentals of nursing course before

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Information Test | 15 minute
  The blood pressure knowledge test consists of 20 questions. The test is multiple choice and the maximum score that can be obtained from the test is 20 by giving 1 point for each correct item.
Self-Managed Learning Skills Scale | 15 minute
  The instrument was developed to measure self- managed learning skilss. The scale consists of 21 items. The scale is in 5-point Likert type. The minimum score that can be obtained from the scale is 21 and the maximum score is 105. A high score from the scale indicates high self-directed learning skills, while a low score indicates low self-directed learning skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khodaei S, Hasanvand S, Gholami M, Mokhayeri Y, Amini M. The effect of the online flipped classroom on self-directed learning readiness and metacognitive awareness in nursing students during the COVID-19 pandemic. BMC Nurs. 2022 Jan 19;21(1):22. doi: 10.1186/s12912-022-00804-6. PMID 35042484
- [Result] Hu R, Gao H, Ye Y, Ni Z, Jiang N, Jiang X. Effectiveness of flipped classrooms in Chinese baccalaureate nursing education: A meta-analysis of randomized controlled trials. Int J Nurs Stud. 2018 Mar;79:94-103. doi: 10.1016/j.ijnurstu.2017.11.012. Epub 2017 Nov 29. PMID 29223013